CLINICAL TRIAL: NCT02332733
Title: Phase II, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Immunogenicity of Two Doses of the LID/NIAID Live-Attenuated Tetravalent Dengue Vaccine, TV003, Administered Six Months Apart, to Healthy Adults, Adolescents, and Children in Thailand
Brief Title: Evaluating the Safety of and Immune Response to a Dengue Vaccine (TV003) in Healthy Adults, Adolescents, and Children in Thailand
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WRAIR 2041
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TV003 Vaccine (Experimental): Participants will receive a single injection of TV003 at Days 0 and 180.
  Interventions: Biological: TV003
- Placebo vaccine for TV003 (Placebo Comparator): Participants will receive a single injection of placebo for TV003 at Days 0 and 180.
  Interventions: Biological: Placebo for TV003

INTERVENTIONS:
Biological: TV003 — 10^3 plaque forming units (PFU) of rDEN1 delta 30, 10^3 PFU of rDEN2/4 delta 30(ME), 10^3 PFU of rDEN3 delta 30/31-7164, and 10^3 PFU of rDEN4 delta 30 to be administered as 0.5 mL by subcutaneous injection in the deltoid region of the upper arm or the thigh in pediatric participants
  Arms: TV003 Vaccine
Biological: Placebo for TV003 — To be administered as 0.5 mL by subcutaneous injection in the deltoid region of the upper arm or the thigh in pediatric participants
  Arms: Placebo vaccine for TV003

SUMMARY:
The purpose of this study is to evaluate the safety of and immune response to two doses of a dengue vaccine (TV003) given 6 months apart to healthy adults, adolescents, and children in Thailand.

DETAILED DESCRIPTION:
Dengue infection is a leading cause of illness and death in the tropics and subtropics. The infection is caused by any one of four types of the dengue virus. This study will evaluate the safety of and immunogenicity to a vaccine (called TV003) against all four types of the dengue virus in healthy adults, adolescents, and children aged 12 months to 50 years in Thailand.

Participants will be enrolled sequentially in four age groups (adults, adolescents, children, and young children), and researchers will evaluate safety data before enrolling each subsequent cohort. Each participant will be in the study for approximately 12 months.

At study entry (Day 0), participants will be randomly assigned to receive either the TV003 vaccine or a placebo vaccine for TV003. All participants will receive two doses of TV003 or placebo-the first dose at study entry (Day 0) and the second dose 6 months later on Day 180. Additional study visits will occur on Days 6, 9, 12, 15, 28, 56, 72, 186, 189, 192, 195, 208, 236, 252, and 360.

All study visits will include a medical history review and a physical exam. Select study visits will also include blood collection and a urine pregnancy test for participants of childbearing potential.

At the vaccination study visits, participants will remain in the clinic for approximately 30 minutes after each vaccination for observation and monitoring. For 20 days after each vaccination, participants will take their temperatures and record any symptoms. Throughout the entire study period, study researchers will monitor participants for suspected dengue infection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participant between the ages of 12 months and 50 years at the time of enrollment into the study
* Residence within the greater Bangkok area for the entire duration of the study period with access to transportation to study site
* Participants and/or their parents/guardians who the investigator believes can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits)
* Participants who will remain available for the duration of the study, approximately 26 weeks post-second vaccination
* Good general health as determined by physical examination, laboratory screening, and review of medical history
* If the participant is a minor, an assent form (for participant age 7-17 years) and informed consent form signed and dated by minor and the participant's parent(s) or legally acceptable representative, respectively. If the participant is 18 years of age or older, an informed consent form signed and dated by the participant (and by an independent witness if required by local regulations)
* If the participant is female, she must be of non-childbearing potential (i.e., either pre-menarcheal, surgically sterilized, or one year post-menopausal), or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (i.e., intrauterine contraceptive device, condom and spermicide combination, oral contraceptives or other equivalent hormonal contraception [e.g., progestin implantable, cutaneous hormonal patch, or injectable contraceptives]) for 30 days prior to vaccination, have a negative pregnancy test prior to vaccination, and must agree to continue such precautions for 60 days after completion of the vaccination series. Any child who begins menarche during the study period must follow the same precautions listed above, from menarche until 60 days after the second vaccine dose.

Exclusion Criteria:

* Pregnant or lactating female or female planning to become pregnant or planning to discontinue abstinence or contraceptive precautions
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, renal, autoimmune, hematologic, or endocrine disease or functional defect, as determined by history, physical examination, or screening tests
* History of any neurological, psychiatric, or behavioral disorder or seizures, with the exception of a single febrile seizure in childhood
* Self-reported or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent, greater than or equal to 0.5 mg/kg/day or 20 mg/day, for more than 2 consecutive weeks within the past 3 months). Inhaled and topical steroids are allowed.
* Body weight less than 10 kg at the time of enrollment
* HIV infection by screening and confirmatory assays, hepatitis C virus (HCV) infection by screening and confirmatory assays, or hepatitis B virus (HBV) infection by hepatitis B surface antigen (HBsAg) screening
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), or platelet count, as defined in this protocol
* History of allergic disease/reaction likely to be exacerbated by any component of the vaccine; or any history of a severe allergic reaction or anaphylaxis
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Planned administration of any vaccine not foreseen by the study protocol, during the period starting from 30 days before each dose of the study vaccine and ending 30 days after each dose; with the exceptions of standard infant and child inactivated vaccines and the inactivated influenza vaccine or the inactivated rabies vaccine (without administration of immunoglobulin) administered to adults or children
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine/placebo or planned use at any time during the study period
* Administration of immunoglobulins and/or blood products within 90 days preceding the first dose or planned administration at any time during the study period, which might interfere with assessment of the immune response
* A planned or anticipated move to a location that will prohibit participating in the trial for the full 12 month duration
* Potential adult participants or parents of potential child participants, who do not have easy access to a fixed or mobile telephone
* Any participant identified as a site employee of the investigator or study clinic, with direct involvement in the proposed study or other studies under the direction of that investigator or study clinic, as well as any family member (i.e., immediate, husband, wife and their children, adopted or natural) of the clinic employees or the investigator

Ages: 12 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 266 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited local and general adverse events (AEs) within the 21-day (Days 0-20) follow-up period after each vaccine dose | Measured through Day 200
  AEs will be summarized by severity and relationship to vaccine by individuals and each group.
Occurrence of unsolicited AEs within the 21-day (Days 0-20) follow-up period after each vaccine dose | Measured through Day 200
  AEs will be summarized by severity and relationship to vaccine by individuals and each group.
Occurrence of serious adverse events (SAEs) throughout the entire study period | Measured through Day 360
Serum plaque reduction neutralization titer 50% (PRNT50) to DENV-1, DENV-2, DENV-3, and DENV-4 viruses for each participant at baseline (Day 0) and Study Days 28, 56, 72, and 180 following each vaccination | Measured through Day 360
  Monovalent, bivalent, trivalent, and tetravalent seropositivity and seroconversion rates will be determined at these time points. Seroconversion will be defined as a 4-fold or greater rise in DENV-1, DENV-2, DENV-3, or DENV-4 neutralizing antibody titers by Day 72 compared with the pre-vaccination titer.

SECONDARY OUTCOMES:
Frequency of viremia of each monovalent component of the vaccine after the first and second doses of vaccine | Measured through Day 360
  The mean peak of viremia, mean day of onset of viremia, and mean duration of viremia of each monovalent component within each age cohort will be calculated.
Quantity of viremia of each monovalent component of the vaccine after the first and second doses of vaccine | Measured through Day 360
  The mean peak of viremia, mean day of onset of viremia, and mean duration of viremia of each monovalent component within each age cohort will be calculated.
Duration of viremia of each monovalent component of the vaccine after the first and second doses of vaccine | Measured through Day 360
  The mean peak of viremia, mean day of onset of viremia, and mean duration of viremia of each monovalent component within each age cohort will be calculated.
Number of vaccinees infected with DENV-1, DENV-2, DENV-3, and DENV-4 | Measured through Day 360
  Defined by recovery of vaccine virus from the blood or serum of a participant and/or seropositivity OR seroconversion to DENV
Duration of the antibody response in recipients of the tetravalent vaccine | Measured through Day 360
  The PRNT50 to DENV-1, DENV-2, DENV-3, and DENV-4 will be determined for all specimens collected on Study Day 180 following each vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Veerachai Watanaveeradej, MD, Principal Investigator — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Phramongkutklao Hospital, Bangkok, Thailand